CLINICAL TRIAL: NCT01802710
Title: Influence of the Combined Psychological and Medical Treatment in the Improvement of Symptoms and Quality of Life in Patients With Functional Dyspepsia
Brief Title: Clinical Improvement and in Quality of Life-Functional Dyspepsia-
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Miren Orive Calzada, Msc, Hospital Galdakao-Usansolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008111005
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Psychogenic Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological support (Experimental): Ten weekly sessions, which the first 8 were in group and the last 2 were individuals. It consists on a) an informational session; b) Beck's cognitive-behavioural therapy; and c) progressive-muscle relaxation according to Jacobson
  Interventions: Behavioral: Psychological support
- No psychological support (Active Comparator): Patients of this group only received the conventional medical treatment, not receiving any psychological support
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Psychological support
  Arms: Psychological support
Other: No intervention
  Arms: No psychological support

SUMMARY:
Functional dyspepsia (FD)is defined as the presence of symptoms thought to originate in the gastroduodenal region with no evidence of structural disease that is likely to explain the symptoms. The cause of this condition is unclear, not being a recognized treatment for it. The conventional treatments for those patients are symptom based. Unfortunately, these medications are not very effective. Patients with FD report poorer health status, mental health, and social functioning than patients with structural gastrointestinal pathology. Our aim is to compare a combined intervention (medical plus psychological intervention) versus conventional intervention (medical intervention)in regard to the health related quality of life, symptomatology, anxiety and depression of those patients. The investigators hypothesized that compared with conventional intervention a combined intervention would yield significantly better short (after treatment) and medium term (six months after treatment) improvement of health related quality of life and symptoms.

DETAILED DESCRIPTION:
Patients were recruited from the digestive services of Galdakao-Usansolo and Basurto hospitals. They were randomly allocated to the control or experimental group. 82 patients were included in the control group and 76 in the experimental group.

Regarding the intervention, the treatment of the control group was a conventional (medical) intervention. It was focused on the most bothersome symptom. Prokinetic (for example cinitapride) or antisecretory agent (for example omeprazole) was prescribed in standard dose. Experimental group received the combined intervention (medical plus psychological intervention). The psychological support consisted of ten weekly sessions, which the first 8 were in group and the last 2 were individuals. In those sessions the patients received a) an information session to increase the patients' knowledge of functional dyspepsia; b) a Beck's cognitive-behavioural therapy focused on modifying the influence of some cognitive issues to gastrointestinal symptoms; c) and progressive-muscle relaxation according to Jacobson, with the aim to provide the ability to relax in certain stress situations. This technique was created for reducing anxiety by alternately tensing and relaxing the muscles.

All the patients completed all the self questionnaires at baseline (t0), at the end of the treatment (T1) and at six months follow up (T2). The health related quality of life was assessed by the Dyspepsia Related Health Scale (DRHS), and anxiety and depression were assessed by the Hospital Anxiety and Depression Scale (HADS). Finally, the subjective clinical improvement was also considered and it was measured by a question about how they feel in regard to the functional dyspepsia, with five alternatively responses (a) Much better, b) quite a lot better, c) somewhat better, d) about the same, e) somewhat worse, f) quite a lot worse, g) much worse).

ELIGIBILITY:
Inclusion Criteria:

* to have chronic upper abdominal symptoms consistent with ROME III criteria for functional dyspepsia
* to have an endoscopy to exclude structural organic causes at the time of the recruitment

Exclusion Criteria:

* to have any organic pathology that could explain the dyspeptic symptoms
* to be using non-steroidal anti-inflammatory drugs (NSAIDs)
* to suffer physical or psychological impairments preventing them from properly completing the questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Manuel Orive, Doctor, Principal Investigator — Basurto University Hospital; Jose Luis Cabriada, Doctor, Study Chair — Hospital Galdakao-Usansolo; Aitor Orive, Doctor, Study Chair — Hospital Galdakao-Usansolo; Begoña Matellanes, Psychology, Study Chair — University of Deusto; Maria Josefa Ulloa, Nurse, Study Chair — Basurto University Hospital; Jesus Angel Padierna, Doctor, Study Chair — Hospital Galdakao-Usansolo; Antonio Escobar, Doctor, Study Chair — Basurto University Hospital; Antonio Bernal, Doctor, Study Chair — Hospital Galdakao-Usansolo
Locations (1):
- Galdakao-Usansolo Hospital, Usansolo, Bizkaia, Spain

REFERENCES:
- [Result] Orive M, Barrio I, Orive VM, Matellanes B, Padierna JA, Cabriada J, Orive A, Escobar A, Quintana JM. A randomized controlled trial of a 10 week group psychotherapeutic treatment added to standard medical treatment in patients with functional dyspepsia. J Psychosom Res. 2015 Jun;78(6):563-8. doi: 10.1016/j.jpsychores.2015.03.003. Epub 2015 Mar 11. PMID 25791668

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychological Support: Ten weekly sessions, which the first 8 were in group and the last 2 were individuals. It consists on a) an informational session; b) Beck's cognitive-behavioural therapy; and c) progressive-muscle relaxation according to Jacobson
  Psychological support + conventional medical treatment
- No Psychological Support: Patients of this group only received the conventional medical treatment, not receiving any psychological support
  Only conventional medical treatment
Period: From T0 to T1
Arm/Group | Psychological Support | No Psychological Support
Started | 76 | 82
Completed | 60 | 72
Not Completed | 16 | 10
Period: From T1 to T2
Arm/Group | Psychological Support | No Psychological Support
Started | 60 | 72
Completed | 58 | 70
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: In certain analyzes we lose some subjects, for example when studying Subjective Clinical Improvement (here we have 60 patients in the experimental group and 69 in the control group)
Groups:
- No Psychological Support: Patients of this group only received the conventional medical treatment, not receiving any psychological support
  No psychological intervention
- Total: Total of all reporting groups
Arm/Group | Psychological Support | No Psychological Support | Total
Number analyzed (Participants) | 76 | 82 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.28 (14.06) | 47.09 (15.19) | 45.73 (14.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 66 | 130
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  Spain | 76 | 82 | 158

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DYSPEPSIA RELATED HEALTH SCALE (DRHS)
Description: The Dyspepsia Related Health Scale (DRHS) is a self-reported dyspepsia-specific questionnaire that consists of four scales: severity of common symptoms, pain intensity, pain disability, and satisfaction with dyspepsia-related health. The score, for each scale, ranges between 0 and 100, with 0 representing the most severe situation and 100 the least severe. It also yields a global score that ranges from 0 to 100, with higher scores indicating less severe dyspepsia. The adapted and validated Spanish version of this questionnaire is known as QoL-PEI (Quality of Life in relation to Stomach and Intestinal Problems Questionnaire). Its reliability was found to be satisfactory (Cronbach's alpha 0.92). Its factorial analysis confirmed the four scales found by the DRHS but added a global score scale. The convergent validity was moderate (0.54).
Time Frame: Participants will be followed at the recruit moment (t0) after treatment (t1) and six months after treatment (t2)
Population: the number analyzed in the rows differs from overall number analyzed because, as it is occur in follow-up studies, patients were lost from T0 to T1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychological Support | No Psychological Support
Number analyzed (Participants) | 76 | 82
units on a scale
  Change from t0 to t1 in DRHS-severity symptoms: number analyzed (Participants) | 60 | 72
  Change from t0 to t1 in DRHS-severity symptoms | 73.72 (16.76) | 65.31 (17.60)
  Change from t0 to t2 in DRHS-severity symptoms: number analyzed (Participants) | 58 | 70
  Change from t0 to t2 in DRHS-severity symptoms | 71.85 (20.46) | 64.89 (19.22)

2. Secondary Outcome: Subjective Clinical Improvement
Description: Subjective clinical improvement was measured by a question about how patients feel in regard to the functional dyspepsia ("In relation to functional dyspepsia, how would you rate your health now? a)much better; b) quite a lot better; c) somewhat better; d) about the same; e) somewhat worse; f) quite a lot worse; g) much worse
Time Frame: Subjective clinical improvement it is measured after treatment (t1) and six months after treatment (t2)
Measure: Count of Participants; unit: Participants
Groups:
- Psychological Support: Ten weekly sessions, which the first 8 were in group and the last 2 were individuals. It consists on a) an informational session; b) Beck's cognitive-behavioural therapy; and c) proressive-muscle relaxation according to Jacobson
  Psychological support + conventional medical treatment
Arm/Group | Psychological Support | No Psychological Support
Number analyzed (Participants) | 60 | 69
Participants
  Better in relation to functional dyspepsia at T1 | 37 | 17
  Better in relation to functional dyspepsia at T2 | 36 | 26

3. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale
Description: It is a 14-item measure: 7 items evaluate depression (the HADS-D subscale) and 7 evaluate anxiety (the HADS-A subscale). For each subscale items range from 0 to 21. A subscale score of 0-7 indicates the absence of anxiety or depression; a score of 8-10 indicates a possible case of anxiety or depression; and a score of 11 or higher indicates the presence of anxiety or depression. It has been adapted and validated in a Spanish population
Time Frame: Participants will be followed at the recruit moment (t0) after treatment (t1) and six months after treatment (t2)
Population: The number analyzed in the rows differs from overall number analyzed because, as it is occur in follow-up studies, patients were lost from T0 to T2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychological Support | No Psychological Support
Number analyzed (Participants) | 76 | 82
units on a scale
  Change From t0 to t1 in HADS-D: number analyzed (Participants) | 72 | 60
  Change From t0 to t1 in HADS-D | 8.95 (1.95) | 9.31 (2.00)
  From t0 to t2in HADS-D: number analyzed (Participants) | 58 | 70
  From t0 to t2in HADS-D | 9.09 (1.88) | 9.71 (2.01)

ADVERSE EVENTS:
Description: "0" Total Number of Participants at Risk: All-Cause Mortality, Serious and other adverse events were not monitored/assessed
Groups:
- Psychological Support: Ten weekly sessions, which the first 8 were in group and the last 2 were individuals. It consists on a) an informational session; b) Beck's cognitive-behavioural therapy; and c) progressive-muscle relaxation according to Jacobson
  Psychological support
- No Psychological Support: Patients of this group only received the conventional medical treatment, not receiving any psychological support
  No intervention
Arm/Group | Psychological Support | No Psychological Support
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes